CLINICAL TRIAL: NCT05466058
Title: Validity of Palpation in Detecting the Site of Lesion in Diabetic Trigger Finger Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eslam Elsayed Ali Shohda (Other Government)
Responsible Party: Sponsor-Investigator, Eslam Elsayed Ali Shohda, Dr - teaching fellow, General Committee of Teaching Hospitals and Institutes, Egypt
Organization: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Eslam Elsayed Ali
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Trigger Finger; Validity of Palpation
Keywords: trigger finger
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Intervention Model Description: case control clinical trial
Who Masked: Investigator
Masking Description: radiologist will not know if the participant has trigger finger or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases (Other): Physical therapist will assess patients to detect site of pathology (A1, A2, A3, A4, A5, midpalm or wrist) then patients will be refereed to radiologist who will detect site of pathology by sonography
  Interventions: Diagnostic Test: palpation - ultrasonography
- control (Other): Physical therapist will assess patients to detect site of pathology (A1, A2, A3, A4, A5, midpalm or wrist) then patients will be refereed to radiologist who will detect site of pathology by sonography
  Interventions: Diagnostic Test: palpation - ultrasonography

INTERVENTIONS:
Diagnostic Test: palpation - ultrasonography — Physical therapist will assess patients to detect site of pathology (A1, A2, A3, A4, A5, midpalm or wrist) then patients will be refereed to radiologist who will detect site of pathology by sonography

SUMMARY:
Aim of the study: 1) to determine validity of palpation in detecting the site of lesion in trigger finger patients by detecting sensitivity specificity, positive and negative predictive values. Hypothesis: Sensitivity of T.F palpation will be ≥ 0.70 and Specificity of T.F palpation will be ≥ 0.70.

DETAILED DESCRIPTION:
Trigger finger (T.F) is a disorder characterized by snapping or locking of a finger. Painful popping or clicking sound is elicited by flexion and extension of the involved digit. It is a multifactorial disease . The common mechanism of triggering is that there is a mismatch of diameter between flexors tendons and the annular pulley (retinacular sheath) of the finger. A1 pulley is the most common site of pathology; hence some authors define T.F generally as a disease of A1 pulley . Many case reports revealed that A2 or A3 pulley is a site of triggering . Others revealed that flexor retinaculum or palmar aponeurosis is the site of pathology. In some cases, after intraoperatively surgeons release A1 pulley they found still triggering and found the triggering at other site . So clinician should examine all possible sites of affection before any topical procedures application or surgery, hence our question is in T.F patients is palpation valid in detecting the site of lesion? Design and Setting: the investigator propose a case control clinical trial to enroll TF patients (cases) and non TF diabetic patients (control) to detect sensitivity specificity, positive and negative predictive values for finger palpation. The study will be conducted in physical therapy outpatient clinic and radiology department at Alahrar teaching hospital, Zagazig, Egypt.

Procedures: Patients will be referred by orthopedist who knows inclusion and exclusion criteria, he will refer 31 cases (patients who agree to participate in this study). Diabetic patients without Tf (155) will by refereed from outpatient clinics (control). Physical therapist will assess patients to detect site of pathology (A1, A2, A3, A4, A5, midpalm or wrist) then patients will be refereed to radiologist who will detect site of pathology by sonography.

ELIGIBILITY:
Inclusion Criteria:

1 - Diabetic patients will be included to this study if they have TF (cases) as clinically evaluated and refereed by orthopedist and diabetic patients not complaining of TF(control).

Exclusion Criteria:

1. patients with complete locked finger.
2. Ages below 18 y is .
3. Patients with any other hand pathology .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
validity of palpation in detecting the site of lesion in trigger finger patients by detecting sensitivity specificity, positive and negative predictive values | 6 month - 1 year
  validity of palpation in detecting the site of lesion in trigger finger patients by detecting sensitivity specificity, positive and negative predictive values

CONTACTS AND LOCATIONS:
Overall Officials: Eslam Elsayed Shohda, phd, pt, Principal Investigator — GOTHI

IPD SHARING:
Plan to Share IPD: Undecided
think about that